CLINICAL TRIAL: NCT07077733
Title: Comparison of Postoperative Sore Throat Following Endotracheal Intubation Performed With Videolaryngoscope, Videostylet, and Fiberoptic Bronchoscope
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ayşe meryem yalçın, anesthesiology resident, Hacettepe University
Other Study IDs: KA-23060
Record Dates: First submitted 2025-06-28; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Sore Throat
Keywords: videolaryngoscope; videostylet; fiberoptic bronchoscope; postoperative sore throat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Video laryngoscopy: Patients who underwent intubation using a videolaryngoscope
- Video stylet: Patients who underwent intubation using a video stylet
- Fiberoptic bronchoscopy: Patients who underwent intubation using fiberoptic bronchoscopy

SUMMARY:
This study aims to compare video laryngoscope (VL), video stylet (VS), and fiberoptic bronchoscope (FOB) in elective endotracheal intubations of patients aged 18 to 65 years, classified as ASA I-II and without predicted difficult airways. The primary endpoints are the incidence of postoperative sore throat and hoarseness, while secondary endpoints include intubation time, first-attempt intubation success, hemodynamic responses, and procedure-related complications. Postoperative sore throat and hoarseness will be assessed at the bedside at the 20th minute and 6th hour following extubation.

DETAILED DESCRIPTION:
Objective: The selection of an appropriate device for endotracheal intubation is essential for successful airway management. Although various publications in the literature compare the techniques used for intubation in terms of their advantages and disadvantages, there remains a lack of consensus regarding the superiority of one method over another. This study aims to compare video laryngoscope (VL), video stylet (VS) and fiberoptic bronchoscope (FOB) devices in patients without anticipated difficult airway undergoing elective intubation, primarily in terms of postoperative sore throat and hoarseness, and secondarily in terms of intubation time, first-attempt success rate, hemodynamic responses, and complications.

Materials and Methods: The study included patients aged 18-65 years, with ASA physical status I-II, who underwent elective surgery under general anesthesia at the operating rooms of Hacettepe University Hospitals, and who had no predictors of a difficult airway. Patients were allocated into three groups: Group VL (n=105) was intubated using the iS3-L Video Laryngoscope (Shenzhen Insighters Medical Technology, Gaung Dong, China); Group VS (n=102) using the iS3-R Video Rigid Stylet (Shenzhen Insighters Medical Technology, Gaung Dong, China); and Group FOB (n=104) using the iS3-C Video Flexible Laryngoscope (Shenzhen Insighters Medical Technology, Gaung Dong, China).

The primary outcome was the incidence of postoperative sore throat and hoarseness at the 20th minute and 6th hour postoperatively. Secondary outcomes included intubation time, first-attempt success rate, hemodynamic responses to intubation, and complications during the procedure.

Sample size calculations were performed using the G*Power 3.1.9.6 (Franz Faul, Universität Kiel, Kiel, Germany) software. To detect at least a 20% difference in the incidence of postoperative sore throat between any two groups with 80% power and a 5% significance level, the required total sample size was calculated as 294 patients. However, accounting for potential exclusions and data loss, a minimum of 102 patients per group was targeted.

This was a non-randomized, comparative clinical study. The anesthesiologist responsible for each case was not interfered with regarding the management of general anesthesia or the method of endotracheal tube insertion.

ELIGIBILITY:
Inclusion Criteria:

* The requirement for endotracheal intubation for general anesthesia during elective surgery in our hospital
* Being between 18 and 65 years of age
* Having an ASA physical status classification of I or II
* Providing informed consent to participate in the study

Exclusion Criteria:

* Presence of a coagulation disorder
* Being identified as a patient with a predicted difficult airway (Patients anticipated to have a difficult airway during standard preoperative anesthesia evaluation and documented as such in the preoperative assessment notes. Relevant criteria include: Mallampati score of 3 or 4, upper lip bite test grade 3, short neck length, abnormal neck anatomy or limited neck mobility, micrognathia/retrognathia, facial deformities/trauma, and mouth opening less than 3 cm.)
* Presence of obesity (body mass index > 35 kg/m²)
* Undergoing head and neck surgery in which postoperative sore throat is expected due to the surgical site
* Placement of a nasogastric (NG) tube during surgery, which may contribute to postoperative sore throat
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 65 years with an ASA physical status score of I or II, who underwent elective surgery under general anesthesia at the operating rooms of Hacettepe University Hospital, were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 311 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
incidence of postoperative sore throat and hoarseness | 6 hours postoperatively
  Primary aim of this study is to compare video laryngoscope (VL), video stylet (VS) and fiberoptic bronchoscope (FOB) devices in patients without anticipated difficult airway undergoing elective intubation, in terms of postoperative sore throat and hoarseness at the 20th minute and 6th hour postoperatively.

SECONDARY OUTCOMES:
intubation time | from the beginning to the end of the intubation procedure
  The duration between the placement of the airway device, selected by the attending anesthesiologist, into the patient's mouth and the confirmation of successful intubation (as indicated by the appearance of end-tidal CO₂ on the capnograph) was recorded as the intubation time.
first-attempt success rate | from the beginning to the end of the intubation procedure
  The success of intubation with the selected airway device on the first attempt was recorded; in cases where the first attempt failed, the total number of intubation attempts was noted.
hemodynamic responses to intubation | from the beginning to the end of the intubation procedure
  The patient's hemodynamic changes during intubation were noted
complications during the intubation | from the beginning to the end of the intubation procedure
  Complications during intubation were noted

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe Üniversitesi, Ankara, altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes